CLINICAL TRIAL: NCT05458583
Title: Comparison of Periodontal Status and Failure Rates With Different Retainer Bonding Methods and Adhesives: A Randomized Clinical Trial
Brief Title: The Periodontal Status and Failure Rates With Different Retainer Bonding Techniques Using One-step Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Serpil Cokakoglu, Assistant Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E-60116787-020-14577
Record Dates: First submitted 2022-06-28; First posted 2022-07-14 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Periodontal Inflammation
Keywords: failure rate; periodontal status; retainer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator who performed the assessment of the periodontal status was blinded to study groups. Moreover, the person performing data entry and the statistician was blinded to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Direct bonding with conventional adhesive (Other): The fixed retainer was applied with direct bonding technique using two-step (conventional) adhesive
  Interventions: Procedure: Baseline periodontal measurements (T0); Procedure: Periodontal measurements (T1); Procedure: Periodontal measurements (T2); Procedure: Retainer failure rates
- Direct bonding with one-step adhesive (Other): The fixed retainer was applied with direct bonding technique using one-step adhesive
  Interventions: Procedure: Baseline periodontal measurements (T0); Procedure: Periodontal measurements (T1); Procedure: Periodontal measurements (T2); Procedure: Retainer failure rates
- Indirect bonding with conventional adhesive (Other): The fixed retainer was applied with indirect bonding technique using two-step (conventional) adhesive
  Interventions: Procedure: Baseline periodontal measurements (T0); Procedure: Periodontal measurements (T1); Procedure: Periodontal measurements (T2); Procedure: Retainer failure rates
- Indirect bonding with one-step adhesive (Other): The fixed retainer was applied with indirect bonding technique using one-step adhesive
  Interventions: Procedure: Baseline periodontal measurements (T0); Procedure: Periodontal measurements (T1); Procedure: Periodontal measurements (T2); Procedure: Retainer failure rates

INTERVENTIONS:
Procedure: Baseline periodontal measurements (T0) — Periodontal measurements including plaque index, gingival index and calculus index were recorded at the bonding session.
Procedure: Periodontal measurements (T1) — Periodontal measurements including plaque index, gingival index and calculus index were recorded at the 6 months after bonding.
Procedure: Periodontal measurements (T2) — Periodontal measurements including plaque index, gingival index and calculus index were recorded at the 12 months after bonding.
Procedure: Retainer failure rates — A retainer with at least one composite pad detachment was considered to be a failure during 1-year follow-up.

SUMMARY:
The aim of this study was to evaluate fixed retainers, bonded with either direct or indirect techniques using one- or two-step adhesives, in terms of periodontal status and failure rates.

ELIGIBILITY:
Inclusion Criteria:

* Good treatment outcomes
* good oral hygiene
* No systemic or periodontal problems
* No extraction or missing anterior teeth and restorations

Exclusion Criteria:

- Patients unwilling to wear a fixed retainer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Plaque index measurements | at the bonding session
  Plaque index was scored by a specialized periodontist on the mesiolingual, lingual, and distolingual sides of each tooth at the bonding session based on the following scale: 0 (no plaque), 1 (a film of plaque adhering to the free gingival margin and adjacent area of the tooth), 2 (moderate accumulation of soft deposits within the gingival pocket, or on the tooth and gingival margin which can be seen with the naked eye) and 3 (abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin).
  All measurements were performed using acrylic stents to ensure reproducible placement of the periodontal probe (PCP 15 UNC, Hu-Friedy, Chicago, IL).
Plaque index measurements | 6 months (T1) after bonding
  Plaque index (PI) was scored by a specialized periodontist on the mesiolingual, lingual, and distolingual sides of each tooth at 6 months after bonding based on the following scale: 0 (no plaque), 1 (a film of plaque adhering to the free gingival margin and adjacent area of the tooth), 2 (moderate accumulation of soft deposits within the gingival pocket, or on the tooth and gingival margin which can be seen with the naked eye) and 3 (abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin).
  All measurements were performed using acrylic stents to ensure reproducible placement of the periodontal probe (PCP 15 UNC, Hu-Friedy, Chicago, IL).
Plaque index measurements | 12 months (T2) after bonding
  Plaque index was scored by a specialized periodontist on the mesiolingual, lingual, and distolingual sides of each tooth at 12 months after bonding based on the following scale: 0 (no plaque), 1 (a film of plaque adhering to the free gingival margin and adjacent area of the tooth), 2 (moderate accumulation of soft deposits within the gingival pocket, or on the tooth and gingival margin which can be seen with the naked eye) and 3 (abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin).
  All measurements were performed using acrylic stents to ensure reproducible placement of the periodontal probe (PCP 15 UNC, Hu-Friedy, Chicago, IL).
Gingival index measurements | at the bonding session
  Gingival index was scored by a specialized periodontist on the mesiolingual, lingual, and distolingual sides of each tooth at bonding session based on the following scale: 0 (absence of inflammation), 1 (mild inflammation), 2 (moderate inflammation) and 3 (severe inflammation).
  All measurements were performed using acrylic stents to ensure reproducible placement of the periodontal probe (PCP 15 UNC, Hu-Friedy, Chicago, IL).
Gingival index measurements | 6 months (T1) after bonding
  Gingival index was scored by a specialized periodontist on the mesiolingual, lingual, and distolingual sides of each tooth at 6 months after bonding based on the following scale: 0 (absence of inflammation), 1 (mild inflammation), 2 (moderate inflammation) and 3 (severe inflammation).
  All measurements were performed using acrylic stents to ensure reproducible placement of the periodontal probe (PCP 15 UNC, Hu-Friedy, Chicago, IL).
Gingival index measurements | 12 months (T2) after bonding
  Gingival index was scored by a specialized periodontist on the mesiolingual, lingual, and distolingual sides of each tooth at 12 months after bonding based on the following scale: 0 (absence of inflammation), 1 (mild inflammation), 2 (moderate inflammation) and 3 (severe inflammation).
  All measurements were performed using acrylic stents to ensure reproducible placement of the periodontal probe (PCP 15 UNC, Hu-Friedy, Chicago, IL).
Calculus index measurements | at bonding session
  Calculus index was scored by a specialized periodontist on the mesiolingual, lingual, and distolingual sides of each tooth at bonding session based on the following scale: 0 (no calculus present), 1 (supragingival calculus covering not more than one third of the exposed tooth surface), 2 (supragingival calculus covering more than one third but not more than two thirds of the exposed tooth surface or the presence of individual flecks of subgingival calculus around the cervical portion of the tooth or both) and 3 (supragingival calculus covering more than two thirds of the exposed tooth surface or a continuous heavy band of subgingival calculus around the cervical portion of the tooth or both).
  All measurements were performed using acrylic stents to ensure reproducible placement of the periodontal probe (PCP 15 UNC, Hu-Friedy, Chicago, IL).
Calculus index measurements | 6 months after bonding
  Calculus index was scored by a specialized periodontist on the mesiolingual, lingual, and distolingual sides of each tooth at 6 months after bonding based on the following scale: 0 (no calculus present), 1 (supragingival calculus covering not more than one third of the exposed tooth surface), 2 (supragingival calculus covering more than one third but not more than two thirds of the exposed tooth surface or the presence of individual flecks of subgingival calculus around the cervical portion of the tooth or both) and 3 (supragingival calculus covering more than two thirds of the exposed tooth surface or a continuous heavy band of subgingival calculus around the cervical portion of the tooth or both).
  All measurements were performed using acrylic stents to ensure reproducible placement of the periodontal probe (PCP 15 UNC, Hu-Friedy, Chicago, IL)
Calculus index measurements | 12 months after bonding
  Calculus index was scored by a specialized periodontist on the mesiolingual, lingual, and distolingual sides of each tooth at 12 months after bonding based on the following scale: 0 (no calculus present), 1 (supragingival calculus covering not more than one third of the exposed tooth surface), 2 (supragingival calculus covering more than one third but not more than two thirds of the exposed tooth surface or the presence of individual flecks of subgingival calculus around the cervical portion of the tooth or both) and 3 (supragingival calculus covering more than two thirds of the exposed tooth surface or a continuous heavy band of subgingival calculus around the cervical portion of the tooth or both).
  All measurements were performed using acrylic stents to ensure reproducible placement of the periodontal probe (PCP 15 UNC, Hu-Friedy, Chicago, IL)

SECONDARY OUTCOMES:
Failure rate | during 1-year follow-up
  A retainer with at least one composite pad detachment was considered to be a failure during a 1-year follow-up period. When there was no wire breakage or deformation, the tooth surfaces were cleaned and bonding was completed using a direct technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Faculty of Dentistry Department of Orthodontics, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No